CLINICAL TRIAL: NCT05858762
Title: Study of an Artificial Intelligence Algorithm for the Classification of Digital Tomosynthesis Breast Images for Automated Breast Cancer Diagnosis
Brief Title: Artificial Intelligence for Automated Diagnosis of Breast Cancer
Acronym: AICAMAMMELLA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS1414/20
Record Dates: First submitted 2023-03-28; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer Diagnosis
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Breast digital tomosynthesis — Introduction of an almost three-dimensional imaging technique called breast digital tomosynthesis

SUMMARY:
Mammography is a two-dimensional imaging technique which involves the tissues overlapping under the projective image; dense glandular tissue above or below the lesion can reduce the visibility of the lesion.

The trouble could be the interpretation of the image obtained which may lead to the inability to visualize a fist stage cancer and the probability that to a healthy person will be diagnosed a pathology that is not present (false positive). The introduction of an almost three-dimensional technique imaging called breast digital tomosynthesis (DBT) can overcome most limitations. In the last 5 years image analysis methods based on Artificial Intelligence (, AI) have also been massively introduced in breast cancer detection. The study is a prospective observational study based on Artificial intelligence whose the mail goal is to develop a method to identify a lesion.

ELIGIBILITY:
Inclusion Criteria:

* Patients who refer to the Regina Elena for diagnostic mammography tests
* Informed consent

Exclusion Criteria:

* presence of prostheses, artifacts, outcomes of a study in the breast intervention under the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing mammography
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Artificial Intelligence system to detect a lesion | 12 months
  Lesion detction is based on breast density, case type, BIRADS assessment categories, mammographic appearance, size and pathological profile of malignant lesions

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Università degli Studi di Napoli Federico II, Napoli
  - "Regina Elena" National Cancer Institute, Rome

IPD SHARING:
Plan to Share IPD: Undecided